CLINICAL TRIAL: NCT03238625
Title: Painless Local Anaesthesia With Bicarbonate Admixture: A Phase II, Monocentric, Double-blind, Randomized, Placebo-controlled Crossover Trial
Brief Title: Painless Local Anaesthesia With Bicarbonate Admixture
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LIDOBICARB
Record Dates: First submitted 2017-06-21; First posted 2017-08-03 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Local Infiltration; Anesthesia
MeSH Terms: interventions — Lidocaine; Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Consisting of 24 individuals between 18 and 75 years, able to understand German, not pregnant, with no intolerance of local anesthetics, with intact skin and no skin diseases, not prone to bleeding or taking anticoagulation or aspirine.
  Intervention: Every individual receives four injections IMP1: Lidocaine and sodium bicarbonate ratio 3:1, IMP 2: Lidocaine and sodium bicarbonate ratio 9:1, IMP 3: Lidocaine, and IMP 4: Sodium cloride 0.9% (=placebo), namely two in every volar forearm, and has to rate the pain associated during the injection of the fluid, not the needle stitch. Afterwards the anesthetic effect on the four areals which got injected will be checked with a palomar laser after 5, 30, 60, 90, 120 and 180 minutes.
  Interventions: Drug: Lidocaine and sodium bicarbonate; Drug: Lidocaine; Drug: Sodium cloride 0.9%
- Group 2 (Placebo Comparator): Consisting of 24 different individuals than those belonging to Group 1. Between 18 and 75 years, able to understand German, not pregnant, with no intolerance of local anesthetics, with intact skin and no skin diseases, not prone to bleeding or taking anticoagulation or aspirine.
  Intervention: Every individual receives two injections:
  IMP 3 Lidocaine, and IMP 4 Sodium cloride 0.9% (=placebo), namely one in every volar forearm, and has to rate the pain associated during the injection of the fluid, not the needle stitch. Afterwards the anesthetic effect on the two areals which got injected will be checked with a palomar laser after 5, 30, 60, 90, 120 and 180 minutes.
  Interventions: Drug: Lidocaine; Drug: Sodium cloride 0.9%

INTERVENTIONS:
Drug: Lidocaine and sodium bicarbonate — Lidocaine and sodium bicarbonate ratio 3:1
  Arms: Group 1
Drug: Lidocaine and sodium bicarbonate — Lidocaine and sodium bicarbonate ratio 9:1
  Arms: Group 1
Drug: Lidocaine — Lidocaine injection
Drug: Sodium cloride 0.9% — Placebo

SUMMARY:
This study examines whether the injection of local anesthesia mixed with sodium bicarbonate in the ratio of 3:1 creates a less burning sensation and is as effective regarding the anesthetic effect as in the ratio of 9:1.

DETAILED DESCRIPTION:
Therefore the investigators compare two groups with 24 healthy individuals in each group in a cross-over study. One group receives four injections (two in each forearm) and one group receives only two injections (one in each forearm)

The four injections of group 1 are:

* IMP1: Lidocaine and sodium bicarbonate ratio 3:1
* IMP 2: Lidocaine and sodium bicarbonate ratio 9:1
* IMP 3: Lidocaine
* IMP 4: Sodium cloride 0.9% (=placebo)

The two injections of group 2 are IMP1 and IMP2.

After each injection the individual has to rate their pain sensation on a NRS scale and afterwards the anesthetic effect gets tested by a standardized laser application.

ELIGIBILITY:
Inclusion Criteria:

* healthy male or female individuals between 18 and 75 years
* able to understand and speak German
* able to follow the instructions

Exclusion criteria:

* oversensitivity to lidocaine or other local anesthetics of amide type or sulfites
* prone to bleeding, intake of aspirine or anticoagulation
* pregnancy
* skin on forearms with lesions (i.e. sunburn, wounds, eczema or other skin diseases)

  * previous participation at the same study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2017-10-18 (Actual)

PRIMARY OUTCOMES:
Rating of injection pain between IMP1 and IMP2 | 1 minute
  on NRS scale

SECONDARY OUTCOMES:
rating of injection pain of IMP3 and IMP4 | 1 minute
  on NRS scale
rating of clinical relevance of the difference between pain sensation of the injections | 5 minutes
  participant can choose between four adjectives regarding injection pain:
  * desirable
  * acceptable
  * less acceptable
  * unacceptable
assessment of local anesthesia of each injection with a standardized laser | 90 minutes
  with Palomoar Synosure non-ablative Fractional CO2-Laser with 30 mJ, 15 ms
duration of anesthetic effect of each injection | maximum 90 minutes
  with Palomoar Synosure non-ablative Fractional CO2-Laser with 30 mJ, 15 ms

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital, Department of Dermatology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No